CLINICAL TRIAL: NCT04066309
Title: Implant Retained Rehabilitation With Surgical and Prosthetic Digital Workflow: A Randomized Clinical Trial
Brief Title: Implant Retained Rehabilitation With Surgical and Prosthetic Digital Workflow
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Neodent (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS.I.001
Record Dates: First submitted 2019-08-19; First posted 2019-08-26 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Jaw, Edentulous, Partially
Keywords: Dental Implants; Bone-Implant Interface; Mouth Rehabilitation
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Intervention Model Description: Two implants (one of each group) will be placed on each subject at the same stage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abutment removal (Experimental): At the time of surgery, customizable healing abutments will be placed on implants. These will be replaced by Pro PEEK Abutments 21 days later to placement of temporary prostheses (loading). The final abutments (Titanium Bases) and final prostheses will be inserted 2 months after loading.
  Interventions: Device: Neodent GM Helix Implant; Device: GM Customizable Healing Abutment; Device: GM Pro PEEK Abutment; Device: GM Exact Titanium Base
- Final abutment (Experimental): The final abutments (Titanium Bases) will be placed at the time of the implant placement surgery and will stay at mouth during all period of the study. Temporary and final prosthesis will be placed on Titanium Bases.
  Interventions: Device: Neodent GM Helix Implant; Device: GM Exact Titanium Base

INTERVENTIONS:
Device: Neodent GM Helix Implant — 4.0x10 mm Neodent GM Helix Implants will be placed 2mm subcrestally (in relation to the buccal bone plate) in the posterior region of the maxilla, under local anesthesia and with adequate bone bed preparation, as recommended by the manufacturer, using the guided surgery technique.
Device: GM Customizable Healing Abutment — Customizable healing abutments will be placed at the time of implant placement.
  Arms: Abutment removal
Device: GM Pro PEEK Abutment — Placement of temporary single prostheses (early loading), over temporary abutments.
  Arms: Abutment removal
Device: GM Exact Titanium Base — Insertion of the final abutment (Titanium Base and Zirconia Coping), following the digital workflow.

SUMMARY:
The aim of this study is to prospectively collect clinical data to confirm the safety and clinical performance of Neodent Titanium Base Abutment and Pro PEEK Abutment in daily dental practice setting, by means of a randomized clinical study of prosthetic rehabilitation using these devices.

A total of 48 healed implant sites (at least 4 months post-extraction) shall be included during the sample enrollment (24 patients), which will be randomly divided into two groups, so that each patient receives one implant from each group (removal and non-removal of the abutment placed at the time of surgery).

Patients will be followed for 24 months after implant loading. It is expected that there is no difference in peri-implant bone level change between the two treatment groups.

DETAILED DESCRIPTION:
The study protocol was reviewed and approved by an Ethics Committee (EC) in Brazil.

Sample size was calculated based on an alpha level of 5% and beta of 20% to detect a mean intergroup difference of 0.2mm, with a standard deviation of 0.2mm, in peri-implant bone level change 24 months after implant loading. Sample size calculation showed that a sample of 17 implants is needed for each group. With rate of 2 implants per patient and a "worst-case" drop-out rate of 20%, a sample size of 24 patients resulting in an estimated number of 24 implants, in each group, is thought to be sufficient to allow statistical analysis of clinical outcome data.

A total of 48 healed implant sites (at least 4 months post-extraction) shall be prospectively and consecutively selected during the sample enrollment (24 patients).

Data concerning the studied variables will be collected in the following stages: Screening (First visit); TP - Implant placement; TT - Impressions for temporary prosthesis confection (2 ± 1 days prior to T0); T0 - Implant Loading (temporary prosthesis placement - 21 ± 1 days after implant placement); TF - Impressions for final prosthesis confection (10 ± 1 business days prior to T6); T2 - Final prosthesis placement (2 months ± 1 week after loading); T12 and T24 - 12 and 24 months ± 1 month, respectively, after loading.

In both study groups, 4.0x10 mm Neodent GM Helix Implants will be placed 2mm subcrestally (in relation to the buccal bone plate) in the posterior region of the maxilla, under local anesthesia and with adequate bone bed preparation, as recommended by the manufacturer, using the guided surgery technique. Two implants (one of each group) will be placed in the same individual, to be restored by single prostheses.

In Group 1, customizable healing abutments will be placed at the time of implant placement. Twenty-one days later, the implants will be loaded by means of placement of temporary single prostheses (early loading), fabricated with centric and eccentric occlusal contacts [1], over temporary abutments (Pro PEEK Abutment). The final prosthesis will be delivered after a 2-months period of implant loading. Thus, digital models will be obtained (intraoral scanning or conventional impression and model scanning) 10 ± 1 business days prior to T2 (TF) for the confection of the final prostheses, to be placed over Titanium Bases and Zirconia Copings, following the digital workflow.

The transgingival height of the Titanium Base shall be selected by the clinician so as to leave, preferably, a distance greater than or equal to 2mm between the cementation line of the Zirconia Coping over the Titanium Base and the cementation line of the prosthesis over the Zirconia Coping due to assure better esthetics of the final prosthesis.

In Group 2, the final abutment will be placed at the time of surgery and will not be replaced during the rehabilitation process. A Titanium Base and a Zirconia Coping will be placed over the implant at TP, without loading (placement of an acrylic cap, without occlusal contact, to cover the coping), planned using the initial intraoral scans. Implants will be restored following the same time interval of Group 1, with temporary prosthesis placement in 21 days after surgery, and with final prosthesis placement 2 months thereafter. The clinician shall evaluate the need to re-prepare the Zirconia Coping edge line before obtaining the digital models (intraoral scanning or conventional impression and model scanning) for prostheses confection, in order to obtain the proper distance between the previously mentioned cementation lines.

In both groups, prostheses' passivity, occlusal and interproximal adjustments shall be checked, to avoid compromising the implant/prosthesis set.

Standardized digital periapical radiographs and close-up view photographs will be taken in an usual daily practice frequency, as determined by the investigator to verify prostheses setting and the osseointegration process. Computed tomography Scans will be obtained, in addition to pre-surgery, at T2 for evaluation of clinical parameters and comparison with the implant position planned by guided surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* 2 upper posterior teeth missing, with adjacent natural tooth;
* Healed implant sites (at least 4 months post-extraction);
* Qualify for placement of 4.0x10 mm Neodent GM Helix implants;
* Adequate bone height to allow the 2mm subcrestal placement of a 10-mm-long implant.

Exclusion Criteria:

As exclusion criteria, solely the device contraindications according to the IFU (instructions for use) will be applied:

* Signs of allergy or hypersensitivity to the chemical ingredients of the materials: titanium, titanium alloy (Ti6Al4V-ELI) or PEEK (Polyetheretherketone);
* Presence of acute inflammatory or infectious processes in live tissue;
* Unsuitable bone volume or quality;
* Serious medical problems (e.g. bone metabolism disorders, blood clotting disorders, unsuitable healing capacity);
* Insufficient oral hygiene;
* Incomplete jawbone growth;
* Patient uncooperative and not motivated;
* Abuse of drugs or alcohol;
* Psychosis;
* Prolonged functional disorders which resist any treatment with medications;
* Xerostomia;
* Weakened immunological system;
* Diseases which require the use of steroids;
* Uncontrolled endocrinological diseases;
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Amount of peri-implant bone level change | 2, 6, 12 and 24 months after implant loading
  Peri-implant bone level will be measured on the periapical radiographs obtained as the distance between the coronal margin of the implant shoulder and the most coronal point of the peri-implant bone, on the mesial and distal surfaces of each implant. The horizontal measurement of the remodeling will be done, when there is no bone contact in the cervical part of the implant. This measurement will be performed from the superior site of the bone crest to the lateral edge of the implant, perpendicular to the long axis of the implant.

SECONDARY OUTCOMES:
Implant survival | 2, 6, 12 and 24 months after implant loading
  Implant survival will be defined as no loss of the implant at each follow-up.
Implant success | 2, 6, 12 and 24 months after implant loading
  Evaluation of implant success will be assessed based on the criteria proposed by Buser et al.
Prosthetic survival | 2, 6, 12 and 24 months after implant loading
  Prosthetic survival will be assessed as the prosthesis remaining in situ at each follow-up, irrespective of its condition.

OTHER OUTCOMES:
Prosthetic success | 2, 6, 12 and 24 months after implant loading
  Success will be defined as the prosthesis that remained unchanged and did not require any intervention, except routine occlusal adjustments, during the entire observational period.
Patient Satisfaction: OHIP-14 (Oral Health Impact Profile) questionnaire | Baseline, 2, 6, 12 and 24 months after implant loading
  The Portuguese translation of OHIP-14 [18,19] questionnaire will be used to assess Oral Health Related Quality of Life (OHRQoL), as a measure of patient satisfaction with treatment. Scores will range from 0 (absence of negative impacts on oral health) to 28 (high frequency of negative impacts on oral health).
Clinician Satisfaction: VAS (Visual Analogue Scale) questionnaire | Baseline, 21 days, 2, 6, 12 and 24 months after implant loading
  The assessment will be performed by means of a questionnaire using a visual analog scale (VAS) in the form of a 10 cm horizontal line, where 0 (left end) indicates minimum satisfaction and 10 (right end) indicates maximum satisfaction. The clinician will be instructed to mark the position considered to best represent their degree of general satisfaction with patient treatment. The score will be measured in centimeters from the left end of the line to the marked point.
Rate of adverse events related to the implant, prosthesis, surgery and oral health | Throughout study, up to 24 months after implant loading
  Determined by patient assessment.
Keratinized Tissue Width | Baseline, 21 days, 2, 6, 12 and 24 months after implant loading
  Probes calibrated at 1, 2, 3, 5, 7, and 10 mm will be used to measure keratinized tissue width as the distance from the gingival margin to the mucogingival junction, at the mid-buccal point.

CONTACTS AND LOCATIONS:
Overall Officials: Larissa Trojan, PhD, Study Chair — Neodent
Locations (1):
- Instituto Latino Americano de Pesquisa e Ensino Odontológico (ILAPEO), Curitiba, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No